CLINICAL TRIAL: NCT01269840
Title: Comparison of Monopolar In-Growth and Loose Bipolar Radial Head Implants in the Treatment of Irreparable Radial Head Fractures
Brief Title: Comparison of Two Radial Head Implants
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Rush University (Other); North Shore University Hospital (Other)
Responsible Party: Principal Investigator, John Berschback, Orthopedic surgeon, Northwestern University
Other Study IDs: STU00008411
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Radial Head Fractures
MeSH Terms: conditions — Radial Head and Neck Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In severe injuries of the radial head with multiple, displaced fracture fragments and concomitant ligament damage, excision of the fragments and replacement of the radial head with a metallic implant are indicated. Current radial head implants are composed of metal or a combination of metal and high molecular weight polyethylene. The prostheses are assembled intra-operatively as a solid unit (monopolar) or as an articulating implant with motion between the stem and head (bi-polar). The stem of the implant is inserted into the proximal radius for support and can be classified as either loose-fitting or fixed. According to the investigators, there are no studies that directly compare the clinical and radiographic outcomes between different radial head implant designs. The purpose of this retrospective study is to compare the clinical and radiographic results in patients treated for an irreparable radial head fracture with either a smooth stem, bipolar radial head implant or a monopolar, in-growth radial head implant. The study findings may provide useful clinical information regarding the similarities and differences in these two implant designs.

DETAILED DESCRIPTION:
Data has been completed.

ELIGIBILITY:
Inclusion Criteria:

* Suffered radial head fracture requiring radial head replacement with the Katalyst or Acumed Radial Head Implant from 2002-2009

Exclusion Criteria:

* Unwilling to provide informed consent
* Traumatic brain injury that occurred at the time of elbow fracture

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering radial head fractures, with or without other elbow injuries, requiring radial head replacement
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2010-03; Primary Completion 2012-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Disability of Arm, Shoulder, and Hand (DASH) | 1 clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: John Berschback, MD, Study Director — Northwestern University
Locations (3):
- United States (3):
  - Northwestern University/Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University/Midwest Orthopaedics at Rush, Chicago, Illinois
  - North Shore University Hospital, Evanston, Illinois